CLINICAL TRIAL: NCT00634231
Title: A Phase I Study of AdV-tk + Prodrug Therapy in Combination With Radiation Therapy for Pediatric Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PeBrTK01; NCT00729105 (obsolete NCT alias)
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Malignant Glioma; Recurrent Ependymoma
Keywords: Malignant glioma; Glioblastoma multiforme; Anaplastic astrocytoma; Recurrent ependymoma; Gene therapy; Immunotherapy
MeSH Terms: conditions — Glioma; Ependymoma; Glioblastoma; Astrocytoma | interventions — Valacyclovir; Prodrugs; Radiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AdV-tk (Experimental): AdV-tk + valacyclovir in combination with standard of care radiation
  Interventions: Biological: AdV-tk; Drug: valacyclovir; Radiation: Radiation

INTERVENTIONS:
Biological: AdV-tk
Drug: valacyclovir
  Other Names: Prodrug
Radiation: Radiation
  Other Names: Radiation therapy

SUMMARY:
This study will evaluate the administration of AdV-tk followed by valacyclovir in children with malignant glioma, including glioblastoma multiforme (GBM) and anaplastic astrocytoma (AA), as well as recurrent ependymomas in combination with radiation therapy. The primary objective is to determine if this approach is safe and can be effectively delivered without disturbing standard therapy.

DETAILED DESCRIPTION:
This is an Open label, Phase I, dose escalation study. Patients will receive an injection of AdV-tk into the tumor or tumor bed during the surgical procedure followed by 14 days of anti-herpetic prodrug, valacyclovir, starting 1-3 days after vector injection. Standard radiotherapy will begin 3-7 days after AdV-tK injection. Standard chemotherapy may begin after completion of valacyclovir at the discretion of the treating physician and family. Two dose levels of AdV-tk will be evaluated with a fixed dose of valacyclovir.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 3 years of age or older
* Patients must be planning to undergo standard of care treatment with surgery and radiation therapy.
* Patients must have malignant glioma or recurrent ependymoma
* Tumor must be accessible for injection and must not be located in the brainstem or deep midbrain
* Performance Score: Karnofsky ≥60% if >10y/o, Lansky ≥60 if ≤10y/o
* Bone Marrow Function: Patients must have adequate bone marrow function defined as a peripheral absolute neutrophil count ≥ 1000/µl, platelet count ≥ 100,000/µl (transfusion independent) and hemoglobin ≥ 8.0 gm/dL
* Renal Function: Patients must have serum creatinine ≤ 1.5 times upper limit of institutional normal for age and/or GFR ≥ 70 mL/min/1.73 m2.
* Hepatic Function: Bilirubin ≤ 1.5 times institutional normal; SGPT (ALT) < 3 times institutional normal
* Serum electrolyte values (sodium, potassium, magnesium, calcium) must be checked prior to enrollment and clinically significant abnormalities corrected prior to surgery/AdV-tk injection
* Patients with seizure disorder may be enrolled if well controlled
* Signed informed consent according to institutional guidelines must be obtained

Exclusion Criteria:

* Prior or ongoing liver disease including known cirrhosis, hepatitis B or C infection but not to exclude patients with a distant history of resolved hepatitis A infection
* Patients on immunosuppressive drugs (with exception of corticosteroid)
* Known history of HIV or underlying immunodeficiency
* Patients with acute infections (viral, bacterial or fungal infections requiring therapy)
* Pregnant or breast-feeding patients. Female patients of childbearing age must have negative serum or urine pregnancy test within 1 week of beginning therapy
* Other serious co-morbid illness or compromised organ function
* No other investigational anti-tumor agents within 30 days prior to study entry or during active participation in the study (defined as from study entry until tumor progression)

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 2 months

SECONDARY OUTCOMES:
Overall survival | 5 years
Progression-free survival | 5 years
Objective tumor response | 5 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago (Formerly Children's Memorial Hospital), Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kieran MW, Goumnerova L, Manley P, Chi SN, Marcus KJ, Manzanera AG, Polanco MLS, Guzik BW, Aguilar-Cordova E, Diaz-Montero CM, DiPatri AJ, Tomita T, Lulla R, Greenspan L, Aguilar LK, Goldman S. Phase I study of gene-mediated cytotoxic immunotherapy with AdV-tk as adjuvant to surgery and radiation for pediatric malignant glioma and recurrent ependymoma. Neuro Oncol. 2019 Mar 18;21(4):537-546. doi: 10.1093/neuonc/noy202. PMID 30883662